CLINICAL TRIAL: NCT01648946
Title: Transfusion Requirements in Critical Clinical Oncologic Patients: a Phase 3 Randomized Controlled Clinical Trial (TRICCOP STUDY)
Brief Title: Transfusion Requirements in Critically Ill Oncologic Patient
Acronym: TRICCOP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Fabricio Sanchez Bergamin, Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSB
Record Dates: First submitted 2012-07-19; First posted 2012-07-25 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Anemia
Keywords: Strategies of transfusion; Red blood cells; Liberal; Restrictive; Oncologic critically ill patients
MeSH Terms: conditions — Anemia | interventions — Erythrocyte Transfusion; Erythrocyte Count; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal Transfusion Strategy (Active Comparator): Red blood cell (RBC) transfusion will be given when hemoglobin falls below 9 g/dL since ICU admission until the discharge of intensive care unit. Following administration of 1 RBC unit, a repetition of hemoglobin levels is performed; if a patient's hemoglobin level is 9 g/dL or higher, no additional transfusion is necessary.
  Interventions: Biological: Red blood cell transfusion
- Restrictive Transfusion Strategy (Active Comparator): Red blood cell (RBC) transfusion will be only given when hemoglobin falls below 7 g/dL since ICU admission until the discharge of intensive care unit. Following administration of 1 RBC unit, a repetition of the hematocrit is performed; if a patient's hemoglobin is 7 g/dL or higher, no additional transfusion is necessary.
  Interventions: Biological: Red blood cell transfusion

INTERVENTIONS:
Biological: Red blood cell transfusion — Red blood cell (RBC) transfusion will be given when hemoglobin falls below 9 g/dL since ICU admission until the discharge of intensive care unit. Following administration of 1 RBC unit, a repetition of hemoglobin levels is performed; if a patient's hemoglobin level is 9 g/dL or higher, no additional transfusion is necessary.
  Other Names: • Red blood cells; • Transfusion; • Liberal; • Oncologic critically ill patient
  Arms: Liberal Transfusion Strategy
Biological: Red blood cell transfusion — Red blood cell (RBC) transfusion will be only given when hemoglobin falls below 7 g/dL since ICU admission until the discharge of intensive care unit. Following administration of 1 RBC unit, a repetition of the hematocrit is performed; if a patient's hemoglobin is 7 g/dL or higher, no additional transfusion is necessary.
  Other Names: • Red blood cells; • Transfusion; • Restrictive; • Oncologic critically ill patient
  Arms: Restrictive Transfusion Strategy

SUMMARY:
Blood transfusion in critical ill patients has been associated to several complications and worse outcome. Particularly in oncologic patients, red blood cell transfusion has been investigated as a factor of worse outcome and cancer recurrence due impairment of cellular immunity. Although red blood cell transfusion has decreased in worldwide clinical practice, this issue still remains a matter of controversy in oncologic patients. There are no prospective studies comparing outcomes between restrictive or liberal blood transfusion strategy in oncologic critical patients. This study is a prospective and randomized study comparing clinical outcomes between two strategies of transfusion in oncologic critical patients - liberal or restrictive.

DETAILED DESCRIPTION:
Blood transfusion is commonly performed in critically ill patients, particularly in oncologic patients. However, there are many studies reporting adverse effects of this intervention and final data on benefits are not available. There are no prospective studies in oncologic patients regarding red blood cell transfusions requirements. There are observational and experimental studies suggesting worse outcomes including higher rates of infection and other clinical complications, maybe higher cancer recurrence, in patients submitted to red blood transfusion. Hemoglobin levels around 9 g/dL are usually recommended although not based in evidence . The investigators purpose is to prospectively evaluate two strategies of transfusion in 400 patients with cancer admitted to intensive care unit for severe clinical condition: a liberal strategy - patients receive blood transfusion when hemoglobin is lower than 9 g/dL since the admission to ICU until ICU discharge; a restrictive strategy - patients receive blood transfusion only when hemoglobin is lower than 7 g/dL.

Clinical outcomes, costs and quality of life will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with cancer admitted to ICU due to severe clinical condition AND
* Septic shock diagnosis AND
* Solid neoplasm AND
* Written informed consent

Exclusion Criteria:

* Age less than 18 years OR
* Leukemia or myelodysplastic syndrome OR
* Hematologic neoplasm OR
* Palliative treatment OR
* Renal Chronic Failure in Renal Replacement Therapy OR
* Karnofsky Status < 50 OR
* Previous thrombocytopenia (platelet number lower than 50.000/mm3) OR
* Previous known coagulopathy OR
* Life-threatening bleeding OR
* Documented wish against transfusion OR
* Patients who refused participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
To compare mortality between groups 28 day after ICU admission | 28 days after ICU admission

SECONDARY OUTCOMES:
To compare length of stay in ICU between groups | 90 days
To compare length of stay in hospital between groups | 90 days
To compare days free of organ dysfunction between groups | 28 days
Adverse effects of transfusion | Followed up until ICU discharge; an expected average of one week
  I. Haemolytic complications after transfusion of RBC; Defined by the clinician on the basis of haemoglobinuria or increased free plasma haemoglobin.
  II. Anaphylactic/allergic reactions; Defined by the clinician on the basis of mucocutaneous signs and symptoms.
  III. Transfusion associated acute lung injury (TRALI); defined as:
  * Acute or worsening hypoxaemia ((PaO2/FiO2 < 40 (PaO2 in kPa) or <300 (PaO2 in mmHg) regardless of PEEP) OR > 50% relative increase in FiO2.
  * Occurrence within 6 hours after RBC transfusion AND
  * Acute or worsening pulmonary infiltrates on frontal chest x-ray OR clinical signs of overt pulmonary oedema.
  IV. Ischaemic events; Defined as either myocardial, cerebral, intestinal or acute limb ischaemia
Mortality | 60 day
  All cause 60 day mortality
All cause 90 day mortality All cause 90 day mortality Mortality | 90 day
  All cause 90 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Paulo G. Hoff, MD, PhD, Study Director — ICESP - HCFMUSP
Locations (1):
- Instituto do Cancer do Estado de Sao Paulo - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836